CLINICAL TRIAL: NCT04286750
Title: Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple-ascending Doses of ACT-1004-1239 in Healthy Subjects
Brief Title: Study in Healthy Subjects to Examine the Safety and Tolerability of ACT-1004-1239 Given as Multiple, Gradually Increasing Doses and to Examine the Effects of ACT-1004-1239 on the Body and the Way the Body Takes up, Distributes, and Gets Rid of ACT-1004-1239
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ID-086-102; 2019-004262-17 (EudraCT Number)
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-1004-1239

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-1004-1239 Dose level 1 (30 mg) to 5 (Experimental): Each dose level will be investigated in a group of 10 male and female subjects (ratio 1:1, male:female), with 8 subjects being administered ACT-1004-239 and 2 subjects matching placebo (ratio 1:1, male:female). Sentinel dosing will be applied at each dose level, i.e., in each group two subjects (ratio 1:1, male:female) will initially receive study treatment (1 on active treatment and 1 on placebo).
  Interventions: Drug: ACT-1004-1239
- Placebo (Placebo Comparator): Each dose level will be investigated in a group of 10 male and female subjects (ratio 1:1, male:female), with 8 subjects being administered ACT-1004-239 and 2 subjects matching placebo (ratio 1:1, male:female). Sentinel dosing will be applied at each dose level, i.e., in each group two subjects (ratio 1:1, male:female) will initially receive study treatment (1 on active treatment and 1 on placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-1004-1239 — ACT-1004-1239 administered as hard capsules for oral use.
  Arms: ACT-1004-1239 Dose level 1 (30 mg) to 5
Drug: Placebo — Matching placebo administered as hard capsules for oral use.
  Arms: Placebo

SUMMARY:
Study in healthy subjects to examine the safety and tolerability of ACT-1004-1239 given as multiple, gradually increasing doses and to examine the effects of ACT-1004-1239 on the body and the way the body takes up, distributes, and gets rid of ACT-1004-1239

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Healthy male or female subject aged between 18 and 55 years (inclusive) at Screening.
* A female subject of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day - 1 and must agree to consistently and correctly use a highly effective method of contraception with a failure rate of ≤1% per year, be sexually inactive, or have a vasectomized partner.
* A female subject of non-childbearing potential must be postmenopausal, or must have a medical history of previous bilateral salpingectomy, bilateral salpingo-oophorectomy, hysterectomy, premature ovarian failure, XY genotype, Turner syndrome, or uterine agenesis.
* A male subject must use adequate contraception from first study treatment administration up to at least 90 days after last administration unless he is vasectomized.
* A male subject must agree to refrain from donation of semen from first study treatment administration up to at least 90 days after last administration.

Exclusion Criteria:

* Previous exposure to ACT-1004-1239.
* Known hypersensitivity to ACT-1004-1239, or any of its excipients.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment.
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the study.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks prior to first study treatment administration.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Pregnant or lactating woman.
* Any cardiac condition or illness that may jeopardize the safety of the study subject per investigator judgment based on medical history or 12-lead ECG measured at Screening.
* Any immunosuppressive treatment within 6 weeks or 5x terminal half-life (t½), whichever is longer, before study treatment administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent (serious) adverse events | From first study treatment administration up to End of Study (EOS). Duration: up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- BlueClinical Phase 1 Hospital de Prelado, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pouzol L, Baumlin N, Sassi A, Tunis M, Marrie J, Vezzali E, Farine H, Mentzel U, Martinic MM. ACT-1004-1239, a first-in-class CXCR7 antagonist with both immunomodulatory and promyelinating effects for the treatment of inflammatory demyelinating diseases. FASEB J. 2021 Mar;35(3):e21431. doi: 10.1096/fj.202002465R. PMID 33595155